CLINICAL TRIAL: NCT02066051
Title: Intense Pulsed Light (IPL) and Meibomian Gland Expression to Treat Ocular Rosacea Secondary to Inactive Chronic Ocular Graft Versus Host Disease (GVHD)
Brief Title: IPL and Meibomian Gland Expression to Treat Ocular Rosacea Ocular GVHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Joanne F. Shen, M.D., Assistant Professor of Ophthalmology, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-003814
Record Dates: First submitted 2014-02-13; First posted 2014-02-19 (Estimated); Results first posted 2015-11-25 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-10

CONDITIONS: GVHD; Ocular Rosacea; Dry Eye Syndrome
MeSH Terms: conditions — Rosacea; Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IPL Treatment (Experimental): Subjects who had inactive chronic graft versus host disease (GVHD) after allogeneic bone marrow transplantation and severe dry eye symptoms related to ocular rosacea unresponsive to conventional management were recruited. Subjects were treated with 4 monthly sessions of intense pulsed light (IPL) and meibomian gland expression.
  Interventions: Device: IPL; Procedure: Meibomian Gland Expression

INTERVENTIONS:
Device: IPL — Intense Pulsed Light (IPL) treatment from Quadra Q4 Platinum Series, made by DermaMed Solutions. With the eyes patched closed the IPL was applied to the surface of the skin by the way of a hand-held wand in 30 spots over the skin in the lower lid, cheek area, and nose area starting and ending from in front of each ear.
Procedure: Meibomian Gland Expression — After the IPL was applied, the eyes were numbed for 15 minutes with a numbing drop, and a sterile cotton swab was used to squeeze the eyelids and express clogged oil secretions from the miebomian glands.

SUMMARY:
The purpose of this study was to see if Intense Pulsed Light (IPL) can be used safely and effectively to help treat dry eyes from ocular rosacea after chronic graft-versus-host disease (GVHD). Current treatment options for this disease are limited.

DETAILED DESCRIPTION:
Ocular rosacea and meibomian gland disease are major contributors to keratoconjunctivitis sicca after chronic GVHD. Rosacea exacerbates the aqueous deficiency caused by damage to lacrimal and accessory lacrimal glands similar to cholestasis damage in the biliary system.

Subjects who had inactive chronic GVHD after allogeneic bone marrow transplantation and severe dry eye symptoms related to ocular rosacea were recruited and treated with 4 monthly sessions of IPL and meibomian gland expression. Their charts were reviewed prior to treatment to confirm quiescence of active systemic disease. Symptom scores were quantified with Ocular Surface Disease Index (OSDI) and Standard Patient Evaluation of Eye Dryness questionnaire (SPEED2). Baseline complete eye exam was performed, and subjects received an eyes assessment score based on the Chronic Graft-Versus-Host Disease (GVHD) Assessment and Scoring Form.

Symptoms, exam, and diagnostic data were obtained at baseline (month 0, month 1, month 2, month 3, month 4, month 5, month 6, month 9 and month 12). IPL treatment and meibomian gland expression was performed at baseline (month 0), month 1, month 2, and month 3.

ELIGIBILITY:
Inclusion Criteria:

* Ocular rosacea with inactive GVHD

Exclusion Criteria:

* Active GVHD
* Facial laser treatment
* Accutane exposure
* Inability to wear sun protection factor (SPF) 30 sunscreen and avoid sun exposure
* Inability to meet study requirements

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Shen, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Arizona, Scottsdale, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Mayo Clinic in Arizona.
Period: Overall Study
Arm/Group | IPL Treatment
Started | 8
Completed | 7
Not Completed | 1
Not completed — Subject developed active GVHD | 1

BASELINE CHARACTERISTICS:
Arm/Group | IPL Treatment
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Responded to Intense Pulsed Light (IPL)
Description: Participants received treatment over 4 months and were monitored for safety and response for an additional 8 months. The symptoms were scored with the Standard Patient Evaluation of Eye Dryness (SPEED2) questionnaire. The SPEED questionnaire presents the four most commonly experienced dry eye symptom groups and asks patients to tick a box for all symptoms that apply to them. The frequency section ratings run from 0 (never) to 3 (constant), and the severity section ratings run from 0 (no problems) to 4 (intolerable), for a total score ranging from 0 (no problem) to 28 (severe problems). Over a 30% improvement in the SPEED2 score equated a response. None of the subjects were expected to get a complete response due to the nature of the damage to their ocular surface from GVHD.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | IPL Treatment
Number analyzed (Participants) | 7
participants
  Participants who responded positively to IPL | 5
  Participants who did not respond to IPL | 2

2. Secondary Outcome: Number of Participants Who Experienced Adverse Events
Description: Participants were screened for any sign of adverse events at each visit by the principal investigator or one of her colleagues.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | IPL Treatment
Number analyzed (Participants) | 7
participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected over 1 year.
Arm/Group | IPL Treatment
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes